CLINICAL TRIAL: NCT05451654
Title: A Prospective, Multicenter, Randomized, Placebo-controlled, Parallel-group, Double-blind Trial to Evaluate the Clinical Efficacy of NanoManganese® on Top of Standard of Care, in Adult Patients With Moderate to Severe Coronavirus Disease 2019 (COVID-19)
Brief Title: NanoMn®_COVID-19 A Prospective, Multicenter, Randomized, Placebo-controlled, Parallel-group, Double-blind Trial to Evaluate the Clinical Efficacy of NanoManganese® on Top of Standard of Care, in Adult Patients With Moderate to Severe Coronavirus Disease 2019 (COVID-19)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the number of patients recruited was not reached because covid cases were low
Sponsor: Medesis Pharma SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020NanoMn-CT01
Record Dates: First submitted 2022-07-07; First posted 2022-07-11 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Drugs, Investigational

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo + SoC (N=30) (Placebo Comparator): This arm is composed by 30 patients.
  * Placebo: administration of 2 mL twice a day (morning and evening) by depositing 1 mL in the gingivo-jugal groove of each cheek with the graduated pipette.
  * Standard of care
  Interventions: Drug: Placebo
- NanoManganese® + SoC (N=90) (Experimental): This arm is composed by 90 patients.
  NanoManganese® + standard of care group:
  * NanoManganese®: administration of 2 mL twice a day (morning and evening) by depositing 1 mL in the gingivo-jugal groove of each cheek with the graduated pipette.
  * Standard of care
  Interventions: Drug: Experimental drug

INTERVENTIONS:
Drug: Placebo — The administration of the treatment consists in a deposit in the gingivo-jugal groove of each cheek with a graduated pipette
  Arms: Placebo + SoC (N=30)
Drug: Experimental drug — The administration of the treatment consists in a deposit in the gingivo-jugal groove of each cheek with a graduated pipette
  Arms: NanoManganese® + SoC (N=90)

SUMMARY:
This is a prospective, multicenter, randomized (3:1), placebo- controlled, parallel-group, double-blind trial.

Patients will be randomized into two arms of treatment:

* Placebo + SoC (N=30)
* NanoManganese® + SoC (N=90)

Patients will be treated and followed-up for 10 days:

* Arterial oxygen partial pressure (PaO2) will be measured at baseline and at days 3, 5 and 10,
* Oxygen saturation, vital signs including respiration rate, pulse rate, blood pressure and body temperature, disease severity (7-point ordinal scale and NEWS2 score) will be measured at baseline and daily,
* Hematology and biochemistry measurements will be done at baseline and at day 3, 5 and 10,
* Pharmacokinetic (Blood Mn concentration) measurements will be done at baseline and at day 3, 5 and 10,
* Biomarkers will be measured at baseline and at day 3, 5 and 10. At the end of the 10-day treatment period, a follow-up visit will be planned between day 15 and day 22. The following.

assessments/examinations will be performed: oxygen saturation, vital signs including respiration rate and body temperature, disease severity (7-point ordinal scale and NEWS2 score), electrocardiogram (ECG), hematology, biochemistry, concomitant therapies, and adverse events.

DETAILED DESCRIPTION:
120 patients will be enrolled in this study, they will be randomly assigned in 2 arms on a 3:1 ratio, 90 patients in the NanoManganese®

+ Standard of Care group and 30 patients in the placebo + Standard of Care group.

This study will be conducted in Brazil and will be conducted in around 8 investigational sites

The investigational products are :

Manganese sulfate monohydrate, MnSO4, H2O (NanoManganese®) will be administered using the microemulsion AONYS® technology. The product is mucoadhesive, it sticks to the mucosa of the cheeks on which it will be deposited and will not be swallowed.

The placebo (Pharmacopoeia soybean oil) will be administered using the same protocol and the same bottle.

Treatments :

NanoManganese® + standard of care group:

* NanoManganese®: administration of 2 mL twice a day (morning and evening) by depositing 1 mL in the gingivo-jugal groove of each cheek with the graduated pipette.
* Standard of care

Placebo + standard of care group:

* Placebo: administration of 2 mL twice a day (morning and evening) by depositing 1 mL in the gingivo-jugal groove of each cheek with the graduated pipette.
* Standard of care The treatments will be administered by the nurse. Duration of treatment: 10 days or until hospital discharge or until death.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patient aged ≥ 18 years
* Patient hospitalized with positive COVID-19, confirmed by a Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) or an antigen test done ≤ 7 days before study entry
* Patient with at least 1 of the National Institutes of Health COVID- 19 clinical symptoms (Fever or chills, Cough, Shortness of breath or difficulty breathing, Fatigue, Muscle or body aches, Headache, New loss of taste or smell, Sore throat, Congestion or runny nose, Nausea or vomiting, Diarrhea) that appeared ≤ 15 days before study entry
* Patient with a peripheral capillary oxygen saturation (SpO2) < 96%, or with an arterial oxygen partial pressure (PaO2) ≤65 mmHg, at study entry
* Female patient of childbearing potential must be willing to use an efficient birth control method during the study and until 3 months after IMP administration.

A woman is considered to be of childbearing potential if she is post menarche, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus, tubal ligation). The following are acceptable contraceptive methods: - Established use of oral, injected, or implanted hormonal methods of contraception - Intrauterine system or placement of an intrauterine device - Double barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam, gel, film, cream, or suppository - True abstinence [periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not acceptable methods of contraception]

* Male patient must be willing to use male contraception (condom) during the study, avoid donating semen during study and until 3 months after last dose of IMP administration.
* Patient must sign the informed consent form
* Patient who have or have not been vaccinated for COVID-19 (1, 2, 3 or 4 shots) can enter the study

Exclusion Criteria:

* Refusal to participate expressed by patient
* Pregnancy or breast-feeding
* Anticipated transfer to another hospital, which is not a study site within 72 hours
* Contraindication to Manganese supplementation
* Patient under Long-term oxygen therapy or invasive ventilation prior to COVID-19 infection
* Patient requiring Continuous Positive Airway Pressure (CPAP), high flow, or Non-Invasive Ventilation (NIV) and a SpO2 <92%
* Patient on invasive mechanical ventilation
* Patient with homozygotic sickle cell disease or methemoglobin.
* Patient receiving a biotherapy as a SoC for COVID-19
* Patient participating in another drug trial
* Patient under guardianship or prisoner
* Patient with a written order for restricted care
* Patient allergic to peanut or soja
* Patient under parenteral nutrition (with Mn in composition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change of the PaO2/FiO2 ratio | 10 days
  Change from baseline to D10 of the PaO2/FiO2 ratio in the NanoManganese® + SoC group and in the placebo+ SoC group.

SECONDARY OUTCOMES:
Proportion of patients with PaO2 > 65 mmHg | 10 days
  Proportion of patients with PaO2 > 65 mmHg at D3, at D5 and at D10, measured preferable after IP administration in the morning.
Change of PaO2 | 10 days
  Change between baseline and D10 of PaO2
Evolution of respiratory rate over time | 10 days
  Evolution of respiratory rate over time
Proportion of patients with SpO2 ≥ 95% | 10 days
  Proportion of patients with SpO2 ≥ 95% at D3, D5 and at D10,
Change of SpO2 | 10 days
  Change between baseline and D10 of SpO2,
Incidence of oxygen use | 10 days
Duration of oxygen use | 10 days
Oxygen free days at D15-22 after inclusion | 10 days
Incidence of noninvasive support (high flow, CPAP, NIV) use | 10 days
Duration of noninvasive support (high flow, CPAP, NIV) use | 10 days
Noninvasive support (high flow, CPAP, NIV) free days during follow- up (between D15 and D22 after inclusion | 10 days
Incidence of invasive mechanical ventilation use, | 10 days
Duration of invasive mechanical ventilation use | 10 days
Invasive mechanical ventilation free days during follow-up (between D15 and D22 after inclusion) | 10 days
Time to improvement of 1 level on seven point ordinal scale | 10 days
  Higher scores indicate a worse outcome
  1. - Not hospitalized, no limitation of activities
  2. - Not hospitalized, limitation of activities
  3. - Hospitalized, not requiring supplemental oxygen
  4. - Hospitalized, requiring supplemental oxygen
  5. - Hospitalized, on non-invasive ventilation or high flow oxygen devices
  6. - Hospitalized, on invasive mechanical ventilation or ECMO
  7. - Death
Clinical status assessed by ordinal scale | 10 days
Proportion of patient transferred in ICU | 10 days
Description of ICU-free days during follow-up (between D15 and D22 after inclusion) | 10 days
Overall survival at day 22 and cause of death | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa BH, Belo Horizonte, Santa Efigenia, Brazil